CLINICAL TRIAL: NCT01586819
Title: Treatment of Lateral Canthal Rhytides With Medium Depth Chemical Peel With or Without Pretreatment With Botulinum Toxin A: A Split-face, Rater-blinded Randomized Control Trial
Brief Title: Lateral Canthal Rhytides With Medium Depth Chemical Peel With or Without Pretreatment With Botulinum Toxin A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Rebecca Tung, Dermatology Division Director, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 203555
Record Dates: First submitted 2011-11-22; First posted 2012-04-27 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Wrinkles
MeSH Terms: interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin (Active Comparator): The botulinum toxin will be injected into the wrinkles. The injections will take about 10 minutes to complete. Five follow-up visits will be scheduled at 1-7 days, 7-10 days, 2.5-3 weeks, and 12-14 weeks.
  Interventions: Drug: Botulinum Toxin
- Chemical Peel Only (Active Comparator): After cleansing the face with a pre-treatment cleansed composed of water and alcohol, the Jessner's peel solution will be applied to the entire face with a large cotton swab. The mixture will be left in place for a few minutes, and then the face will be wiped clean with water. Next, the TCA peel will be applied around the eyes. After leaving in place for a few minutes, cool, iced washcloths will be applied and the face will be wiped clean with water.
  Wound care regimen will consist of dilute acetic acid and either Aquaphor or petroleum jelly.
  Interventions: Procedure: Chemical Peel Only

INTERVENTIONS:
Drug: Botulinum Toxin — The botulinum toxin will be injected into the wrinkles "crow's feet". The injections will take about 10 minutes to complete.
  Other Names: Botox
  Arms: Botulinum Toxin
Procedure: Chemical Peel Only — After cleansing the face with a pre-treatment cleansed composed of water and alcohol, the Jessner's peel solution [a combination of resorcinol (14g), salicylic acid (14g), and lactic acid (85%) in ethanol (95%)] will be applied to the entire face with a large cotton swab. The mixture will be left in place for a few minutes, and then the face will be wiped clean with water. Next, the TCA peel [35% Trichloroacetic acid] will be applied around the eyes. After leaving in place for a few minutes, cool, iced washcloths will be applied and the face will be wiped clean with water. Wound care regimen will consist of dilute acetic acid and either Aquaphor or petroleum jelly.
  Other Names: Jessner's peel solution; TCA peel
  Arms: Chemical Peel Only

SUMMARY:
This study is being done to find out if the use of botulinum toxin prior to a medium strength combination chemical peel (Jessner's peel followed by 35% Trichloroacetic acid peel) will improve the appearance of crow's feet wrinkles when compared to a chemical peel alone. Botulinum toxin type A is a purified substance, derived from a bacteria that block muscular nerve signals. Jessner's Peel, a combination of resorcinol (14g), salicylic acid (14g), and lactic acid (85%) in ethanol (95%), is a superficial chemical peel. These two products/procedures have been FDA approved to improve the appearance of facial wrinkles.

DETAILED DESCRIPTION:
Wrinkling in the skin is caused by habitual facial expressions, aging, sun damage, smoking, poor hydration, and various other factors. There are two major types of wrinkles-dynamic and static. Dynamic wrinkles, which are due to excessive muscle activity, usually of the face, tend to disappear when you relax your facial muscles. The most common of these dynamic wrinkles are frown lines, forehead wrinkles, and eye wrinkles (or crow's feet). However, if the excessive muscle activity is carried on for too long, these do not disappear completely on relaxation, and are thus called static wrinkles. Static wrinkles are formed either by chronic excessive muscle activity or are due to the effects of age and gravity, with a loss of subcutaneous fat. Examples of static wrinkles are the nasolabial folds, which are the deep grooves running from the sides of the nose to the corners of the mouth.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 75 years old
* In good health
* Has static and dynamic lateral canthal wrinkles ("crow's feet")
* Has the willingness and the ability to understand and provide informed consent and communicate with the investigator

Exclusion Criteria:

* Pregnant or lactating
* Has received the following treatments:

  * botulinum toxin injections in the past 6 months
  * ablative laser procedure in the past 6 months
  * radiofrequency device treatment in the past 6 months
  * ultrasound device treatment in the past 6 months
  * medium to deep chemical peel in the past 6 months
  * temporary soft tissue augmentation material in the past year
  * semi-permanent soft tissue augmentation material in the past 2 years
  * permanent soft tissue augmentation material
* Is planning to receive within the next 3 months, any cosmetic procedure (such as any chemical peels, botulinum toxin injections, ablative or non-ablative laser procedures, filler injections, radiofrequency procedures, dermabrasion, ultrasound and face lifting procedures)
* Has an active infection on their face (excluding mild acne
* Has a history of neuromuscular disorders
* Has an allergy to albumin
* Has an allergy to Aquaphor AND petroleum jelly
* Has a history of bleeding disorders
* Is unable to understand the protocol or to give informed consent
* Has a mental illness

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Tung, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola Dermatology, La Grange Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin | Chemical Peel Only
Started | 12 | 14
Completed | 11 | 14
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin | Chemical Peel Only | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.3 (4.8) | 51.9 (7.1) | 49.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Posttreament Results of Chemical Peel if Botox A is Added as Pre-treatment
Description: The primary objective of this study is to determine if pre-treating the orbicularis oculi muscles with botulinum toxin A improves the results of medium depth chemical peels when treating lateral canthal rhytides. The primary dependent variable is the four-point Facial Wrinkle Severity Scale (FWSS): Grade 0 = no wrinkles; Grade 1 = mild wrinkles; Grade 2 = moderate wrinkles; and Grade 3 = severe wrinkles.
Time Frame: Baseline and 12 weeks
Population: Twenty-six female subjects ages 30 to 75 years old were enrolled in this study.
Measure: Median (Inter-Quartile Range); unit: Units on a wrinkle severity scale
Arm/Group | Botulinum Toxin | Chemical Peel Only
Number analyzed (Participants) | 11 | 14
Units on a wrinkle severity scale | 1 [0 to 1] | 2 [1 to 2]
Statistical Analysis 1: Comparison: Chemical Peel Only; The null hypothesis was that subjects receiving Botox A as an added pre-treatment would have lower scores on the facial wrinkle severity scale post-treatment; Test type: Superiority; p = .002, Wilcoxon (Mann-Whitney); Z score = -3.3902

2. Primary Outcome: Change From Pre- to Post-treatment Scores of Chemical Peel if Botox A is Added as Pre-treatment
Description: The primary objective of this study is to determine if there is a significant difference between the change from pre- to post-treatment scores on the facial wrinkle severity scale between the chemical peel control group and the chemical peel plus Botox A treatment group. The primary dependent variable is the four-point Facial Wrinkle Severity Scale (FWSS): Grade 0 = no wrinkles; Grade 1 = mild wrinkles; Grade 2 = moderate wrinkles; and Grade 3 = severe wrinkles.
Time Frame: Baseline and 12 weeks
Population: Twenty-six female subjects ages 30 to 75 years old were enrolled in this study.
Measure: Median (Inter-Quartile Range); unit: Units on a wrinkle severity scale
Arm/Group | Botulinum Toxin | Chemical Peel Only
Number analyzed (Participants) | 11 | 14
Units on a wrinkle severity scale | 2 [2 to 2] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Chemical Peel Only; The null hypothesis was that subjects receiving Botox A as an added pre-treatment would have higher difference scores, pre- to post-treatment, on the facial wrinkle severity scale suggesting a more pronounced effect of the chemical peel in combination with the Botox A therapy; Test type: Superiority; p = .001, Wilcoxon (Mann-Whitney); Z score = 3.6115

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for all patients over the entire analysis period, from baseline to 8-10 weeks following pre-treatment.
Arm/Group | Botulinum Toxin | Chemical Peel Only
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 0/11 | 0/14

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to disclose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes